CLINICAL TRIAL: NCT03513406
Title: Comparison of Reversal of Neuromuscular Blockade With Sugammadex Versus Neostigmine Plus Glycopyrolate in Patients Undergoing Burn Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00141829
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Burns
Keywords: muscle function
MeSH Terms: conditions — Burns | interventions — Sugammadex; Neostigmine; Glycopyrrolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sugammadex (Active Comparator): Muscle relaxant reversal will be attained with sugammadex 2 mg/kgm IV.
  Interventions: Drug: Sugammadex
- Neostigmine (Active Comparator): Muscle relaxant reversal will be attained with neostigmine 50 mcg/kgm plus glycopyrrolate10 mcg/kgm IV.
  Interventions: Drug: Neostigmine; Drug: Glycopyrrolate

INTERVENTIONS:
Drug: Sugammadex — Sugammadex is indicated for the reversal of neuromuscular blockade.
  Arms: Sugammadex
Drug: Neostigmine — Neostigmine is indicated for the reversal of neuromuscular blockade.
  Arms: Neostigmine
Drug: Glycopyrrolate — Glycopyrrolate is used in conjunction with neostigmine to prevent neostigmine's muscarinic effects.
  Arms: Neostigmine

SUMMARY:
The purpose of this study is to learn if there is a difference in recovery time when using sugammadex versus neostigmine. The researchers also hope to add further knowledge and data to the safety of using sugammadex in burn patients who are hypermetabolic.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing burn surgery under general anesthesia

Exclusion Criteria:

* Patients without a non-burned upper extremity
* Renal insufficiency or failure
* Sensitivity or hypersensitivity reaction to sugammadex
* Liver impairment, neuromuscular degenerative disease or dependence on drugs or alcohol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Time to return to a 90% Train of Four (TOF) neuromuscular twitch | Within 24 hours after surgery

SECONDARY OUTCOMES:
Time to endotracheal extubation | Within 24 hours after surgery
Time to discharge from the operating room | Within 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Kovac, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States